CLINICAL TRIAL: NCT00666380
Title: Phase 1a Open-label Dose Escalation Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of the Candidate Plasmodium Falciparum Malaria Protein 010 (FMP010) Administered Intramuscularly With GSK Biologicals' Adjuvant AS01B in Healthy Malaria-Naïve Adults
Brief Title: A Study to Determine the Effects of an Investigational Malaria Vaccine Given to Adults Living in the United States and Thereafter to Adults Living in Kenya
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: GlaxoSmithKline (Industry); United States Agency for International Development (USAID) (U.S. Federal Agency); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); Kenya Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A-14620.a; A-14620 (HSRRB); WRAIR 1417 (Other: Walter Reed Army Institute of Research)
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Malaria
Keywords: Malaria; Vaccine; MSP-1 (merozoite surface protein-1); Phase 1
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 10 ug of FMP010 antigen in 0.5 mL AS01B adjuvant (Experimental)
  Interventions: Biological: Plasmodium falciparum Malaria Protein 010 (FMP010)
- 50 ug of FMP010 antigen in 0.5 mL AS01B adjuvant (Experimental)
  Interventions: Biological: Plasmodium falciparum Malaria Protein 010 (FMP010)

INTERVENTIONS:
Biological: Plasmodium falciparum Malaria Protein 010 (FMP010) — Vaccine antigen is a recombinant protein based on merozoite surface protein-1 (MSP-1) of FVO strain of Plasmodium falciparum, and adjuvant AS01B is a proprietary adjuvant of GSK

SUMMARY:
The purpose of this study is to determine whether an investigational malaria vaccine is safe and induces an immune response against malaria when tested in adults living in the United States.

DETAILED DESCRIPTION:
The study begins with the US phase in which 26 volunteers aged 18 to 50 years will be enrolled to receive an investigational malaria vaccine. The vaccine is made of a malaria protein FMP010 mixed in the adjuvant AS01B. Since this vaccine has not yet been in humans, first, 5 volunteers will get a small (10 µg) dose of FMP010 in AS01B. If it is safe, then 20 volunteers will get 50 µg FMP010 in AS01B. Vaccinations are given IM in the deltoid of the non-dominant arm, every month for 3 months. After each vaccination, the subjects will follow up at clinical trials for evaluation of any adverse events. There will be blood draws to assess safety of the vaccine as well as the level of immune response generated to the vaccine.

Upon receipt of preliminary safety results, the Kenya phase begins in which 30 volunteers who are randomized to receive either 50 µg FMP010 in AS01B (20) or the rabies vaccine (10). Vaccination and is on the same schedule as in the US phase and follow-up is for 112 days.

ELIGIBILITY:
Inclusion Criteria:

* A male or non-pregnant, non-lactating female 18 to 50 years of age (inclusive) at the time of screening
* Free of significant health problems as established by medical history and clinical examination before entering into the study
* Available to participate for duration of study (approximately seven months)
* If the subject is female, she must be of non-childbearing potential (either surgically sterilized or one year post-menopausal) or, if of childbearing potential, she must be capable of preventing pregnancy, have a negative pregnancy test at the time of each vaccination, and must agree to continue such precautions for two months after completion of the vaccination series.
* If the volunteer indicates he/she is active duty military (on the DCT sign-in page and intake form), approval from their supervisor through the Division Director using the Statement of Supervisor's Approval Form must be signed and on file prior to receipt of any test product
* Written informed consent must be obtained from the subject before screening procedures.
* Test of Understanding
* Prior to entry into this study, subjects must score at least 80% correct on a 10- question multiple-choice quiz that assesses their understanding of this study. If they do not score 80% on the initial quiz, the protocol information will be reviewed with them to ensure comprehension, and they will have the opportunity to retest. If a volunteer fails to correctly answer 8 of 10 questions after two attempts they will be excluded from the study.

Exclusion Criteria:

* Prior receipt of any investigational malaria vaccine
* Prior receipt of a vaccine containing either QS-21, MPL or AS02 or AS01
* Use of any investigational or non-registered drug or vaccine other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period
* Administration of chronic (defined as more than 14 days) immunosuppressants or other immune-modifying drugs within six months of vaccination. For corticosteroids, this is defined as prednisone, or equivalent, 0.5 mg/kg/day. Inhaled and topical steroids are allowed.
* Planned administration of a vaccine not foreseen by the study protocol within 30 days of the first dose of the study vaccine
* Any past history of malaria
* Planned travel to malarious areas during the study period
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection
* A family history of congenital or hereditary immunodeficiency
* Chronic or active neurologic disease including seizure disorder
* History of splenectomy
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or abnormal baseline laboratory screening tests

  1. ALT above normal range
  2. Creatinine above normal range
  3. Hemoglobin below normal range
  4. Platelet count below normal range
  5. Total white cell count below normal range
* Acute disease at the time of enrollment (acute disease is defined as the presence of a moderate or severe illness with or without fever). All vaccines can be administered to persons with a minor illness, such as diarrhea or mild upper respiratory infection without fever, i.e., Oral temperature < 37.5°C.
* Hepatomegaly, right upper quadrant abdominal pain or tenderness
* Seropositive for HIV, Hepatitis C virus (antibodies to HCV) and/or HBsAg
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period
* Pregnant or lactating female
* Suspected or known current alcohol abuse/drug abuse as obtained by history and physical examination
* Female who is willing or intends to become pregnant during the study
* Any history of allergic reaction or anaphylaxis to previous vaccination
* Inability to make follow-up visits or complete diary cards
* Allergy to kanamycin, nickel, or imidazole
* Any other significant finding that in the opinion of the investigator would increase the risk of having an adverse outcome from participating in this study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2008-04; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Number of solicited adverse events | 7 days
  Occurrence and intensity of solicited symptoms on day of vaccination and Days 1-7 after each vaccination
Number of unsolicited adverse events | 30 days
  Occurrence and intensity of unsolicited symptoms over a 30-day follow-up period (day of vaccination and 29 subsequent days) after each vaccination
Number of serious adverse events | 1 year

SECONDARY OUTCOMES:
Percent parasite growth inhibition | Up to 112 days
  Functionality of antibodies elicited as measured by percent parasite growth inhibition in GIA against homologous (FVO) and heterologous (3D7) parasites

CONTACTS AND LOCATIONS:
Overall Officials: Michele D Spring, MD, M.S.P.H., Principal Investigator — Walter Reed Army Institute of Research (WRAIR); Nekoye N. Otsyula, M.B. Ch. B., Principal Investigator — Kenya Medical Research Institute
Locations (2):
- Department of Clinical Trials, WRAIR, Silver Spring, Maryland, United States
- USAMRU-K/ KEMRI. Walter Reed Project, Kombewa, Kisumu, Nyanza Province, Kenya

REFERENCES:
- [Derived] Bashir IM, Otsyula N, Awinda G, Spring M, Schneider P, Waitumbi JN. Comparison of PfHRP-2/pLDH ELISA, qPCR and microscopy for the detection of plasmodium events and prediction of sick visits during a malaria vaccine study. PLoS One. 2013;8(3):e56828. doi: 10.1371/journal.pone.0056828. Epub 2013 Mar 15. PMID 23554856
- [Derived] Otsyula N, Angov E, Bergmann-Leitner E, Koech M, Khan F, Bennett J, Otieno L, Cummings J, Andagalu B, Tosh D, Waitumbi J, Richie N, Shi M, Miller L, Otieno W, Otieno GA, Ware L, House B, Godeaux O, Dubois MC, Ogutu B, Ballou WR, Soisson L, Diggs C, Cohen J, Polhemus M, Heppner DG Jr, Ockenhouse CF, Spring MD. Results from tandem Phase 1 studies evaluating the safety, reactogenicity and immunogenicity of the vaccine candidate antigen Plasmodium falciparum FVO merozoite surface protein-1 (MSP1(42)) administered intramuscularly with adjuvant system AS01. Malar J. 2013 Jan 23;12:29. doi: 10.1186/1475-2875-12-29. PMID 23342996